CLINICAL TRIAL: NCT06572488
Title: Exploring the Effects of Non-ablative Er:YAG Laser on Patients Suffering From Recurrent Vulvovaginal Candidiasis
Brief Title: Non-ablative Er:YAG for Recurrent Candidiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espacio Gaspar Clinic (Other)
Responsible Party: Principal Investigator, Adrian Gaspar, Medical Director, Espacio Gaspar Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAND/01
Record Dates: First submitted 2024-08-19; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Candidiasis, Vulvovaginal; Candidiasis of Vagina; Candidiasis, Genital; Recurrent Candidiasis of Vagina; Infection, Candida; Vaginal Yeast Infections
Keywords: non-ablative; Er:YAG laser; Recurrent vaginal yeast infection; Recurrent vulvovaginal candidiasis; candidiasis; vaginal; genital
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Candidiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active therapy with non-ablative Er:YAG laser (Experimental): Patients underwent four laser sessions with non-ablative SMOOTH Er:YAG laser therapy, with 1 moth interval between sessions
  Interventions: Device: Non-ablative SMOOTH mode Er:YAG laser

INTERVENTIONS:
Device: Non-ablative SMOOTH mode Er:YAG laser — Four intravaginal treatments within four months.
  Other Names: SMOOTH mode; non-ablative Er:YAG laser

SUMMARY:
The objective of the study wa to assess the safety, acceptability and effectiveness of non-ablative Er:YAG laser therapy for treatment of symptoms and microbiological conditions of women with recurrent vulvovaginal candidiasis (RVVC). Eligible patients have received 4 laser therapies within four moths and will be assessed at baseline, 3 months and 9 months after last laser therapy.

The effects of laser therapy have been assessed by following the vaginal microbial status, by assessing the five bothersome symptoms related to vaginal infection (burning, itching, dyspareunia, dysuria, and abnormal discharge), by assessing the overall patient satisfaction, and throughout the study the safety of the laser therapy has been monitored.

DETAILED DESCRIPTION:
Genital candidiasis is a common fungal infection that affects both men and women, though it is more frequently observed in women. It is estimated that up to 75% of women will experience at least one episode of vulvovaginal candidiasis (VVC) during their lifetime. The primary causative agents are Candida albicans and other non-albicans pathogenic fungal species.

The likelihood of developing genital candidiasis can be influenced by factors such as age and hormonal changes. Women of reproductive age, especially those who are pregnant, using hormonal contraceptives, or experiencing hormonal fluctuations, are at higher risk. The highest prevalence rate, 9%, is reported among women aged 25 to 34 years. Antibiotic use, which can disrupt the body's microbial balance, is a known risk factor for genital candidiasis, along with other factors like obesity, uncontrolled diabetes, corticosteroid use, chronic stress, and certain lifestyle choices.

Clinical guidelines recommend oral fluconazole or itraconazole as the first-line treatment for recurrent vulvovaginal candidiasis (RVVC). However, after stopping maintenance therapy, a recurrence rate of 40%-50% is expected. While clinical resistance to antifungal agents is rare, overexposure to azoles can lead to resistant strains of C. albicans. Additionally, non-albicans Candida species, such as C. glabrata, often show dose-dependent susceptibility or resistance to fluconazole and other azole agents, and their prevalence is increasing. Given the limited therapeutic options, innovative treatment strategies are necessary.

ELIGIBILITY:
Inclusion Criteria:

* adult women (> 18 years)
* diagnosis of recurrent vaginal yeast infection (> 4 infection per year)

Exclusion Criteria:

* patients having contraindications to laser therapy (epilepsy, pregnancy, acute systemic infection)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Improvement of bothersome symptoms (burning sensation,/irritation, itching or soreness, dyspareunia, dysuria, abnormal vaginal discharge | Change from Baseline at 3 and 9 months after last intervention
  Patients were required to assess the symptom severity on a 0-10 VAS (Visual Analog Pain) scale, 0 referring to "absence of symptom" and 10 referring to "intolerable symptom"

SECONDARY OUTCOMES:
Change in lab cultures of vaginal swabs | Change from Baseline at 3 and 9 months after last intervention
  Lab cultures of vaginal secretion on Sabouraud dextrose agar (SDA) were performed for diagnosis and determination of lead pathogen.
Recording of frequency and severity of adverse effects related to laser treatment | 9 months
  Each visit included recording of any adverse effect. Patients were instructed to report and adverse effect that may have occured during the whole duration of the study.
Patient satisfaction with 5-point Likert scale | Improvement from Baseline at 3 and 9 months after last intervention
  Patients were asked to assess their global satisfaction with the treatment on a 5-point Likert scale (1-Very unsatisfied, 2-Unsatisfied, 3-Neutral, 4-Satisfied, 5-Very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Gaspar, MD, Principal Investigator — Espacio Gaspar Clinic
Locations (1):
- Uroclinica, Mendoza, Argentina

IPD SHARING:
Plan to Share IPD: No